CLINICAL TRIAL: NCT06757374
Title: Evaluation of First-Trimester Maternal Serum Resistin in Hyperemesis Gravidarum
Brief Title: First Trimester Resistin Levels in HG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Mete Kırlangıç, Assoc Prof, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09.2020.1141
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Hyperemesis Gravidarum - Severe; Resistin; Gestational Diabetes Mellitus (GDM)
Keywords: First trimester; maternal serum resistin; hyperemesis gravidarum; HG; GDM
MeSH Terms: conditions — Diabetes, Gestational; Hyperemesis Gravidarum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mild HG (Experimental): In pregnant women admitted in the first trimester, blood samples were first taken and the PUQE-24 questionnaire was used to evaluate the severity of HG, and those with a score of ≤6 were considered as mild HG
  Interventions: Diagnostic Test: Resistin
- Modarete HG (Experimental): In pregnant women admitted in the first trimester, blood samples were first taken and the PUQE-24 questionnaire was used to evaluate the severity of HG, and those with a score of 7-12 were considered as modarete HG
  Interventions: Diagnostic Test: Resistin
- Severe HG (Experimental): In pregnant women admitted in the first trimester, blood samples were first taken and the PUQE-24 questionnaire was used to assess the severity of HG, and those with a score of ≥13 were considered to have severe HG.
  Interventions: Diagnostic Test: Resistin

INTERVENTIONS:
Diagnostic Test: Resistin — Considering the HG effect on endocrinologic and metabolic complications, resistin levels in maternal serum may change in the presence of HG severity
  Other Names: Adipose tissue-specific secretory factor

SUMMARY:
This cross-sectional case-control study was conducted in Tuzla State Hospital Obstetrics Clinic in Turkey. The study evaluated 400 pregnant women during their first trimester of pregnancy. Many pregnant women (50-90%) experience nausea and vomiting during their first trimester; however, some patients have a disease called "hyperemesis gravidarum" (HG) characterized by very severe nausea and vomiting that may require hospitalization. resistin" is a peptide which is secreted primarily by human adipocytes and mononuclear cells. Evidence suggests that resistin increases plasma glucose concentration, reduces glucose intake by adipocytes, and promotes insulin resistance. Considering the HG effect on endocrinologic and metabolic complications, we hypothesized that resistin levels in maternal serum may change in the presence of HG; therefore, the aim of the present study was to evaluate these resistin levels during the first trimester and their correlation with HG severity.

ELIGIBILITY:
Inclusion Criteria:

Those who applied in the first trimester and had a mid-trimester OGTT result

Exclusion Criteria:

1) multifetal pregnancy, 2) fetal chromosomal or structural anomalies, 3) pregestational DM, 4) chronic hypertension or history of preeclampsia, 5) thyroid disease, 5) chronic kidney disease, 6) autoimmune disease, or 7) long-term use of aspirin or glucocorticoids 8) without OGTT results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
PUQE | Immediately after admission in the first trimester
  the PUQE-24 questionnaire was used to evaluate the severity of HG, and those with a score of ≤6 were considered as mild HG, 6-12 as moderate HG, and ≥13 as severe HG

SECONDARY OUTCOMES:
Resistin levels | Immediately after admission in the first trimester
  Resistin levels rise with HG severity
OGTT | admission in 24-28 th week in pregnancy
  After 75 grams of solution was given, blood glucose values were evaluated again at 1st and 2nd hours. GDM was diagnosed when one of the 3 levels of blood sugar was reached or exceeded (Fasting: 92 mg/dl, 1 hour later: 180 mg/dl, 2 hours later: 153 mg/dl).

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lutfi Kirdar City Hospital, Kartal, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddiqui K, George TP. Resistin role in development of gestational diabetes mellitus. Biomark Med. 2017 Jul;11(7):579-586. doi: 10.2217/bmm-2017-0013. Epub 2017 Jul 7. PMID 28685604
- [Background] Vitoratos N, Deliveliotou A, Dimitrakaki A, Hassiakos D, Panoulis C, Deligeoroglou E, Creatsas GK. Maternal serum resistin concentrations in gestational diabetes mellitus and normal pregnancies. J Obstet Gynaecol Res. 2011 Feb;37(2):112-8. doi: 10.1111/j.1447-0756.2010.01327.x. Epub 2010 Dec 16. PMID 21159034
- [Background] Nanda S, Poon LC, Muhaisen M, Acosta IC, Nicolaides KH. Maternal serum resistin at 11 to 13 weeks' gestation in normal and pathological pregnancies. Metabolism. 2012 May;61(5):699-705. doi: 10.1016/j.metabol.2011.10.006. Epub 2011 Dec 5. PMID 22146093